CLINICAL TRIAL: NCT07378904
Title: Intradermal Sterile Water Injection Versus Intravenous Morphine for Renal Colic: A Randomized Controlled Trial
Brief Title: Sterile Water Injection vs Morphine for Renal Colic
Acronym: ISWI-Morph
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Sami Chebbi, Dr, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTHEC-2026-02
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Renal Colic; Urolithiasis
Keywords: Renal Colic; Urinary Stones; Intradermal Sterile Water Injection; Intravenous Morphine; Pain Management
MeSH Terms: conditions — Renal Colic; Urolithiasis; Urinary Calculi; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1:1 ratio to one of three groups: single intradermal sterile water injection (ISWI), four ISWI injections, or intravenous morphine. Each participant will receive only the assigned intervention, and outcomes (pain reduction, analgesic use, patient satisfaction) will be compared between groups. The study is conducted in a double-blind manner, meaning the emergency physician assessing pain and the epidemiologist performing data analysis are blinded to treatment allocation, while patients are aware of the treatment they receive.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Intradermal Sterile Water Injection (1 ISWI) (Experimental): Participants receive 0.5 ml of sterile water injected intradermally at the point of maximal pain in the thoraco-lumbar region (T11-L4). Pain relief is assessed at 5, 30, 45, and 90 minutes.
  Interventions: Procedure: Single Intradermal Sterile Water Injection
- Multiple Intradermal Sterile Water Injections (4 ISWI) (Experimental): Participants receive 1 ml of sterile water divided into four intradermal injections of 0.25 ml each, spaced around the point of maximal pain in the thoraco-lumbar region (T11-L4). Pain relief is assessed at 5, 30, 45, and 90 minutes.
  Interventions: Procedure: Multiple Intradermal Sterile Water Injections
- Intravenous Morphine (Active Comparator): Participants receive intravenous morphine at a dose of 0.1 mg/kg, administered according to local emergency protocols. Pain relief is assessed at 5, 30, 45, and 90 minutes.
  Interventions: Drug: Intravenous Morphine

INTERVENTIONS:
Procedure: Single Intradermal Sterile Water Injection — single 0.5 ml sterile water injection is administered intradermally at the point of maximal pain in the thoraco-lumbar region (T11-L4). Pain will be assessed at 5, 30, 45, and 90 minutes.
  Arms: Single Intradermal Sterile Water Injection (1 ISWI)
Procedure: Multiple Intradermal Sterile Water Injections — 1 ml sterile water is divided into four intradermal injections of 0.25 ml each, spaced around the point of maximal pain in the thoraco-lumbar region (T11-L4). Pain will be assessed at 5, 30, 45, and 90 minutes.
  Arms: Multiple Intradermal Sterile Water Injections (4 ISWI)
Drug: Intravenous Morphine — Morphine is administered intravenously at 0.1 mg/kg according to local emergency protocols. Pain will be assessed at 5, 30, 45, and 90 minutes.
  Arms: Intravenous Morphine

SUMMARY:
This study aims to compare intradermal sterile water injections (ISWI) with intravenous morphine for pain relief in adults with acute renal colic caused by urinary stones. Renal colic is a common emergency characterized by sudden, severe flank pain. Rapid and effective pain control is critical for proper diagnosis and treatment.

Traditional pain management uses NSAIDs or opioids like morphine, which can cause side effects or be limited in certain patients. ISWI is a simple, low-cost, non-systemic method that may provide rapid pain relief by stimulating skin nerves, which can reduce pain signals in the spinal cord and brain.

In this randomized, controlled, double-blind trial, adult patients with confirmed renal stones and pain ≥4/10 on the visual analog scale (VAS) will be assigned to one of three groups:

1. Single ISWI injection
2. Four ISWI injections
3. Intravenous morphine

Pain will be measured at 5, 30, 45, and 90 minutes after treatment. The main goal is to determine whether ISWI is not inferior to morphine in reducing pain at 30 minutes. Secondary goals include comparing the speed and intensity of pain relief between one versus four injections, the need for additional pain medication, and patient satisfaction.

All patients will be monitored for safety, and adverse effects will be recorded. The study follows strict ethical guidelines, including informed consent.

If successful, ISWI could provide a safe, effective, and easily available alternative to morphine for rapid pain relief in renal colic, with minimal side effects, and guide the best injection strategy for optimal patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Acute renal colic with pain score ≥ 4 on the Visual Analog Scale (VAS)
* Urolithiasis confirmed by low-dose abdominopelvic CT scan
* Ability to provide written informed consent

Exclusion Criteria:

* Absence of urinary stones on imaging
* Known allergy or contraindication to morphine or sterile water injection
* Severe renal failure
* Local skin infection at the injection site
* Pregnancy or breastfeeding
* Inability to understand the study or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction at 30 Minutes (VAS) | 30 minutes after intervention
  Change in pain intensity measured using the Visual Analog Scale (VAS) from baseline (before intervention) to 30 minutes after treatment. A decrease of ≥2 points on the VAS is considered effective analgesia.

SECONDARY OUTCOMES:
Pain Reduction at Other Time Points (VAS) | 5, 45, and 90 minutes after intervention
  Proportion of participants requiring additional pain medication during the 90-minute observation period after the assigned intervention.
Need for Rescue Analgesics | 5, 30, 45, and 90 minutes after intervention
  Proportion of participants requiring additional pain medication during the 5, 30, 45, and 90 minutes observation period after the assigned intervention.
Patient Satisfaction | 90 minutes after intervention
  Patient-reported satisfaction with pain management, measured on a 5-point Likert scale at the end of observation (90 minutes).
Adverse Events | 5, 30, 45, and 90 minutes after intervention
  All treatment-related adverse events, including injection site pain, nausea, hypotension, or other complications, monitored at 5, 30, 45, and 90 minutes post-intervention.

OTHER OUTCOMES:
Comparison of Analgesic Effect: Single vs Four ISWI | 5, 30, 45, and 90 minutes after intervention
  Change in pain intensity (VAS) at 5, 30, 45, and 90 minutes comparing participants receiving a single intradermal sterile water injection (0.5 ml) versus four injections (0.25 ml each, total 1 ml). This assesses whether multiple injections provide faster or greater pain relief than a single injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Habib Thameur Teaching Hospital, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Golcuk Y, Demir A, Yildirim B, Acar E. Intradermal sterile water injection in acute renal colic. Am J Emerg Med. 2021 Feb;40:204. doi: 10.1016/j.ajem.2020.05.060. Epub 2020 May 25. No abstract available. PMID 32571630
- [Result] Perros I, Sokhal BS, Swift C, Kitchen M, Mallen C, Somani B. Sterile water injections for analgesia in renal colic: a meta-analysis of level 1 evidence. World J Urol. 2025 Sep 16;43(1):557. doi: 10.1007/s00345-025-05920-x. PMID 40956348
- [Result] Aykanat MC, Kilic M, Cimilli Ozturk T, Ustaalioglu I, Ak R. The efficacy of intradermal sterile water application in severe renal colic: a randomised clinical trial. Urolithiasis. 2023 Oct 12;51(1):121. doi: 10.1007/s00240-023-01496-6. PMID 37823931
- [Result] Moussa M, Papatsoris AG, Chakra MA. Intradermal sterile water injection versus diclofenac sodium in acute renal colic pain: A randomized controlled trial. Am J Emerg Med. 2021 Jun;44:395-400. doi: 10.1016/j.ajem.2020.04.079. Epub 2020 Apr 29. PMID 32444296